CLINICAL TRIAL: NCT01745900
Title: An Evaluation and Comparison of Noninvasive Blood Glucose Concentrations Relative to Finger Capillary Blood Glucose References
Brief Title: Evaluation and Comparison of Noninvasive Blood Glucose Concentrations
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: VeraLight, Inc. (Industry)
Collaborators: InLight Solutions (Industry)
Responsible Party: Sponsor
Other Study IDs: VL-240
Record Dates: First submitted 2012-12-04; First posted 2012-12-10 (Estimated); Last update posted 2012-12-10 (Estimated); Status verified 2012-12

CONDITIONS: Insulin Dependent Diabetes; Non Insulin Dependent Diabetes; Gestational Diabetes
Keywords: Diabetes; Gestational Diabetes; Female
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Diabetes, Gestational; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Comparison of noninvasive glucose measurement performance versus standard invasive reference measurements.

DETAILED DESCRIPTION:
The objectives of this study are

* collect subject data on a near-infrared spectroscopy-based glucose meter
* evaluate existing instrumentation, calibration algorithms and calibration maintenance techniques
* collect data on the physiological and environmental sources of interference and degradation of measurement accuracy.

ELIGIBILITY:
Inclusion Criteria:

* Female aged ≥ 18 and ≤ 50 years of age at time of enrollment
* Females with self reported diagnosis of Type I, Type II or Gestational Diabetes, or no self reported diagnosis of diabetes.

Exclusion Criteria:

* Severe heart disease as evidenced by peripheral edema (self reported)
* Currently taking Lasix (self reported)
* Liver disease as evidenced by jaundice (self reported)
* Receiving dialysis or having known renal compromise (self reported)
* Skin damage at optical sampling site
* Scars, tattoos, rashes or other disruption/discoloration on the right index finger
* Recent (within past month) or current oral steroid therapy or topical steroids applied to the hands; inhaled steroid therapy (self reported)
* Current chemotherapy, or chemotherapy within the past 12 months (self reported)

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Females 18-50 years of age selected from the community 30% with no history of Diabetes 70% with diagnosis of Type I, Type II or Gestational Diabetes
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2012-12; Primary Completion 2013-03 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Continuing validation of near infrared spectroscopy-based glucose meter algorithm | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Amber Brassfield, RN, Principal Investigator — Accelovance
Locations (1):
- Accelovance Inc., San Diego, California, United States